CLINICAL TRIAL: NCT00309738
Title: Study of Pitavastatin Vs. Simvastatin (Following Up-Titration) in Patients With Primary Hypercholesterolemia or Combined Dyslipidemia and 2 or More Risk Factors for Coronary Heart Disease
Brief Title: Study to Compare the Efficacy and Safety of Pitavastatin and Simvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Neil Hounslow, Kowa Research Europe
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NK-104-304
Record Dates: First submitted 2005-12-08; First posted 2006-04-03 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: Kowa; KRE; Hypercholesterolemia; combined dyslipidemia; dyslipidemia; pitavastatin; NK-104; simvastatin
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — pitavastatin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin 4 mg QD (Experimental): Pitavastatin 4 mg once daily
  Interventions: Drug: pitavastatin
- Simvastatin 40 mg QD (Active Comparator): Simvastatin 40 mg once daily
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: pitavastatin
  Arms: Pitavastatin 4 mg QD
Drug: simvastatin
  Arms: Simvastatin 40 mg QD

SUMMARY:
The purpose of this study is to compare the efficacy and safety of pitavastatin with that of simvastatin in patients with risk factors for heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (18-75 years of age)
* At least two cardiovascular disease risk factors
* Must have been following a restrictive diet
* Diagnosis of primary hypercholesterolemia or combined dyslipidemia

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* Conditions which may cause secondary dyslipidemia
* Uncontrolled diabetes mellitus
* Abnormal pancreatic, liver or renal function
* Abnormal serum creatine kinase (CK) above the pre-specified level

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, Med Dr., Study Director — Medical Director
Locations (35):
- Denmark (6):
  - CCBR A/S, Aalborg
  - CCBR A/S, Ballerup Municipality
  - Y Forskning, Bispebjerg Hospital, Copenhagen NV
  - Frederiks Hospital, Kardiologisk, Frederiksberg
  - Kolesterollaboratoriet, Hellerup
  - CCBR A/S, Vejle
- Netherlands (8):
  - Middellaan 5, Breda
  - Bomanshof 8, Eindhoven
  - Damsterdiep 9, Groningen
  - Doezastraat 1, Leiden
  - Kamerlingh Onnesstraat 16-18, Nijmegen
  - Mathenesserlaan 247, Rotterdam
  - Reigerstraat 30, Velp
  - Parkdreef 142, Zoetermeer
- Spain (10):
  - Hospital Clinico S. Juan de Alicante, San Juan, Alicante
  - Hospital Clinic i Provincial, Villaroel, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital de Sagunto, Valencia
- Sweden (11):
  - Angelholms Sjukhus, Medicinkliniken, Angelhom
  - Sahlgrenska University Hospital, Intermedicin, Gothenburg
  - Hjartmottagningen, Helsingborg
  - Lakarcentrum Nyponet, Karineholm
  - Medicinkliniken, Ludvika
  - Hjartmottagningen, Malmo
  - Huslakaren i Sandviken, Sandviken
  - Narsjukhuset Sandviken, Kardiologlab, Medicin, Sandviken
  - Hjart & Karlcenter, Södertälje
  - Karolinska Universitetssjukhuset, Stockholm
  - Hjarthuset AB, Varberg

REFERENCES:
- [Derived] Eriksson M, Budinski D, Hounslow N. Comparative efficacy of pitavastatin and simvastatin in high-risk patients: a randomized controlled trial. Adv Ther. 2011 Sep;28(9):811-23. doi: 10.1007/s12325-011-0056-7. Epub 2011 Aug 25. PMID 21874538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from September 2005 to October 2006 at 43 investigator sites.
Pre-assignment Details: Patients who qualified entered a 6-8 week wash-out/dietary lead-in period followed by a 12- week treatment period. Patients were randomly assigned to one of the two treatment groups: pitavastatin 4 mg QD, or simvastatin 40 mg QD in a ratio of 2:1.
Period: Overall Study
Arm/Group | Pitavastatin 4 mg QD | Simvastatin 40 mg QD
Started | 236 | 119
Safety Population | 233 (Subjects who received at least one dose of study medication) | 119 (Subjects who received at least one dose of study medication)
Completed | 223 | 107
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 4 mg QD | Simvastatin 40 mg QD | Total
Number analyzed (Participants) | 233 | 119 | 352
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 184 | 88 | 272
  >=65 years | 49 | 31 | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (6.82) | 60.9 (6.78) | 60.3 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 37 | 112
  Male | 158 | 82 | 240

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C
Description: Percent change from baseline in low density lipoprotein-cholesterol (LDL-C)
Time Frame: 12 weeks
Population: Subjects who completed the treatment period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pitavastatin 4 mg QD | Simvastatin 40 mg QD
Number analyzed (Participants) | 223 | 107
mg/dL | -43.96 (12.770) | -43.77 (14.416)

2. Secondary Outcome: Number of Patients Attaining NCEP LDL-C Target (< 160 mg/dL)
Description: Number of patients attaining LDL-C target according to National Cholesterol Education Program (NCEP) criteria (< 160 mg/dL)
Time Frame: 12 weeks
Population: Full analysis set (FAS)
Measure: Number; unit: participants
Arm/Group | Pitavastatin 4 mg QD | Simvastatin 40 mg QD
Number analyzed (Participants) | 233 | 118
participants | 203 | 101

ADVERSE EVENTS:
Arm/Group | Pitavastatin 4 mg QD | Simvastatin 40 mg QD
Serious Adverse Events (participants affected / at risk) | 4 | 5
Other Adverse Events (participants affected / at risk) | 51 | 13
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pitavastatin 4 mg QD | Simvastatin 40 mg QD
Lymphadenopathy (Blood and lymphatic system disorders) | 0/233 | 1/119
Acute coronary syndrome (Cardiac disorders) | 1/233 | 0/119
Myocardial infarction (Cardiac disorders) | 1/233 | 0/119
Gastritis (Gastrointestinal disorders) | 1/233 | 0/119
cholelithiasis (Hepatobiliary disorders) | 0/233 | 1/119
Cystitis (Infections and infestations) | 0/233 | 1/119
peritonsilar abscess (Infections and infestations) | 1/233 | 0/119
Syncope (Nervous system disorders) | 0/233 | 1/119
Aortic aneurysm (Vascular disorders) | 0/233 | 1/119
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pitavastatin 4 mg QD | Simvastatin 40 mg QD
Consitpation (Gastrointestinal disorders) | 10/233 | 2/119
Myalgia (Musculoskeletal and connective tissue disorders) | 7/233 | 5/119
Nasopharyngitis (Infections and infestations) | 11/233 | 3/119
Headache (Nervous system disorders) | 13/233 | 3/119
Hypertension (Vascular disorders) | 10/233 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days